CLINICAL TRIAL: NCT01623895
Title: Pharmacogenetic Study in Patients Received Iron Chelating Agent
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyoung Jin Kang, MD. Ph D., Professor, Seoul National University Hospital
Other Study IDs: SNUCH-R-0701
Record Dates: First submitted 2012-06-12; First posted 2012-06-20 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2013-12

CONDITIONS: Hemosiderosis
MeSH Terms: conditions — Hemosiderosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Candidate genes exhibit polymorphisms and encodes proteins that are involved in the pharmacokinetics and pharmacodynamics of deferasirox.
  Candidate genes : MRP2, BCRP, UGT1A subfamily
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate effect of genetic variations on the toxicities and find optimal target population, the investigators planned to analyze the genetic polymorphisms of UDP-glucuronosyltransferase.

DETAILED DESCRIPTION:
Transfusion-associated iron overload induces systemic toxicity. Recently, deferasirox, a convenient long acting oral agent, has been introduced in clinical practice with promising efficacy. However, some patients experience drug-related toxicities and cannot tolerate it. To investigate effect of genetic variations on the toxicities and find optimal target population, we planned to analyze the genetic polymorphisms of UDP-glucuronosyltransferase 1A (UGT1A) subfamily, multi-drug resistance-associated protein 2 (MRP2) and breast cancer resistance protein (BCRP) among pediatric patients received deferasirox.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received deferasirox because of transfusion associated iron overload (Transfusion associated iron overload was defined as ferritin ≥ 1,000 ng/mL in patients who needed over 8 units of RBC transfusions per a year).
2. Patients with written informed consents

Exclusion Criteria:

Patients or parents refusal

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who received deferasirox because of transfusion associated iron overload
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Genetic polymorphism associated with side effects of deferasirox | up to 1 year
  Genetic polymorphism associated with side effects of deferasirox
  - Side effects:
  Increased AST or ALT > 5 x ULN or increased bilirubin > 3 x ULN which was thought to be caused by deferasirox Serum creatinine level increase > 50% above the baseline value.
  * Biospecimen Retention: Samples With DNA
  * Candidate genes exhibit polymorphisms and encodes proteins that are involved in the pharmacokinetics and pharmacodynamics of deferasirox.
  Candidate genes : MRP2, BCRP, UGT1A subfamily

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea